CLINICAL TRIAL: NCT02176733
Title: Trial of Cyclosporine in the Acute Phase of Leber Hereditary Optic Neuropathy
Acronym: CICLO-NOHL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 2010-05
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-01

CONDITIONS: Leber Hereditary Optic Neuropathy
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — Cyclosporine

ARMS (1):
- cyclosporine (Experimental)
  Interventions: Drug: cyclosporine

INTERVENTIONS:
Drug: cyclosporine

SUMMARY:
The Leber Hereditary Optic Neuropathy is a genetic disorder caused by maternal transmission of mitochondrial DesoxiroboNucleid Acid mutations. It is manifested by a rapidly progressive blindness, profound, due to atrophic optic nerve. The visual loss is primarily unilateral bilateralisation taking place in the vast majority of cases in weeks or months. The neuro-cardio-protective properties of cyclosporine (and its analogs specifically targeting the anti-apoptotic mechanisms) are particularly promising.

The investigators hypothesis is that cyclosporine may limit apoptosis during the acute phase of the disease process and would limit the loss of visual acuity and improve the visual prognosis of these patients.

ELIGIBILITY:
Inclusion Criteria:

* patient with the mutation confirmed by molecular analysis
* patient with a recent loss of monocular vision (≤ 6 months)
* voluntarily Patient Consent

Exclusion Criteria:

* patient who have not given their written and informed consent signed
* against indication of cyclosporine
* no drug compliance to previous inclusion
* no national health insurance affiliation
* pregnant women or lactating
* women who could become pregnant during the study period and with no contraception
* private patients of their liberty by judicial or administrative decision, or patients under supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of visual acuity with Monoyer, Early Treatment Diabetic Retinopathy Study and Parinaud scales | at 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Angers, France

REFERENCES:
- [Derived] Leruez S, Verny C, Bonneau D, Procaccio V, Lenaers G, Amati-Bonneau P, Reynier P, Scherer C, Prundean A, Orssaud C, Zanlonghi X, Rougier MB, Tilikete C, Milea D. Cyclosporine A does not prevent second-eye involvement in Leber's hereditary optic neuropathy. Orphanet J Rare Dis. 2018 Feb 17;13(1):33. doi: 10.1186/s13023-018-0773-y. PMID 29454364